CLINICAL TRIAL: NCT00901797
Title: Arthroscopic Rotator Interval Closure in Shoulder Instability Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. maman Eran, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr. Maman
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2009-05

CONDITIONS: Recurrent Shoulder Dislocations
Keywords: ABD; ABDuction; ABR; Arthroscopic Bankart Repair; ACJ; AcromioClavicular Joint; AD; Anterior Drawer; ARIC; Arthroscopic Rotator Interval Closure; BL; Bankart Lesion; CHL; CoracoHumeral Ligament; ER; External Rotation; FF; Forward Flexion; GHJ; GlenoHumeral Joint; HSL; HillSacs Lesion; IR; Internal Rotation; ISP; InfraSPinatus; PD; Posterior Drawer; RI; Rotator Interval; ROM; Range Of Motion; SGHL; Superior GlenoHumeral Ligament; SSC; SubSCapularis; SSP; SupraSPinatus
MeSH Terms: conditions — Shoulder Dislocation; Bankart Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthroscopic Bankart repair (Active Comparator)
  Interventions: Procedure: Arthroscopic Bankart repair
- ABR+ARIC (Active Comparator)
  Interventions: Procedure: ABR+ARIC

INTERVENTIONS:
Procedure: Arthroscopic Bankart repair — Seated in a beach chair position, arm fixed with a skin traction device (Spider shoulder Immobilizer or 3kg traction), arthroscopy through a posterior portal, anterior portal used for inspection and instrumentation, labral lesion released using a suture liberator, full radius and VAPER. Preparation of the glenoid with rasp up and down. Insertion of anchors as necessary into the glenoid and ligation of labral lesion with the sutures. Wound closure with ethilon 4/0 suture, striped dressing, velpeau arm sling.
  Arms: Arthroscopic Bankart repair
Procedure: ABR+ARIC — Seated in a beach chair position, arm fixed with a skin traction device (Spider shoulder Immobilizer or 3kg traction), arthroscopy through a posterior portal, anterior portal used for inspection and instrumentation, labral lesion released using a suture liberator, full radius and VAPER. Preparation of the glenoid with rasp up and down. Insertion of anchors as necessary into the glenoid and ligation of labral lesion with the sutures. Through additional anterior superior portal a suture is passed inferior and adjacent to the SSP and through the superior portion of the Sub Scapularis tendon while the arm in 30 degree of external rotation. Tightening the suture on top of the capsule underneath the deltoid. Wound closure with ethilon 4/0 suture, striped dressing, velpeau arm sling.
  Arms: ABR+ARIC

SUMMARY:
Study Title: Arthroscopic rotator interval closure in shoulder instability repair - a prospective study

Objective: To evaluate the effect of arthroscopic rotator interval closure (ARIC) on patients with recurrent shoulder dislocations undergoing arthroscopic bankart repair (ABR) in terms of recurrence, rehabilitation and function.

Hypothesis:

1. Although Hyperlax patients undergoing ABR have higher incidence of recurrent shoulder dislocations than those without hyperlaxity, adding ARIC will lower the recurrent dislocation rate.
2. Patients with arthroscopic bankart repair (ABR) and ARIC are slower in gaining the range of motion (ROM) but within 6 months are equal to those with ABR only.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-40 years old
* Anterior Shoulder instability
* Hyperlaxity (general and shoulder laxity)

Exclusion Criteria:

* Previous humerus/glenoid fracture
* large bony "Bankart"
* Previous shoulder operation
* Adhesive capsulitis-Habitual dislocations

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Recurrent shoulder dislocation or instability symptoms | Patients will be followed in hospital shoulder clinic 6, 12, 26, 52 weeks post op and then in 1 year intervals until final follow up.

SECONDARY OUTCOMES:
Post operative range of motion (ROM) | Patients will be followed in hospital shoulder clinic 6, 12, 26, 52 weeks post op and then in 1 year intervals until final follow up.
Activity level | Patients will be followed in hospital shoulder clinic 6, 12, 26, 52 weeks post op and then in 1 year intervals until final follow up.
Need for recurrent surgery | Patients will be followed in hospital shoulder clinic 6, 12, 26, 52 weeks post op and then in 1 year intervals until final follow up.
Pain | Patients will be followed in hospital shoulder clinic 6, 12, 26, 52 weeks post op and then in 1 year intervals until final follow up.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Shoulder Unit, Orthopedics B Department, Tel Aviv medical center, Tel Aviv
  - TelAviv Suraski Medical Center, Tel Aviv

REFERENCES:
- [Background] Stokes DA, Savoie FH 3rd, Field LD, Ramsey JR. Arthroscopic repair of anterior glenohumeral instability and rotator interval lesions. Orthop Clin North Am. 2003 Oct;34(4):529-38. doi: 10.1016/s0030-5898(03)00091-9. PMID 14984192
- [Background] Provencher MT, Mologne TS, Hongo M, Zhao K, Tasto JP, An KN. Arthroscopic versus open rotator interval closure: biomechanical evaluation of stability and motion. Arthroscopy. 2007 Jun;23(6):583-92. doi: 10.1016/j.arthro.2007.01.010. PMID 17560472